CLINICAL TRIAL: NCT06495801
Title: Työntekijöiden Sosiaalisen Hyvinvoinnin lisääminen Mobiilisovelluksen Avulla (Effectiveness of a Mobile Application in Improving Employees' Social Well-being)
Brief Title: Effectiveness of a Mobile Application in Improving Employees' Social Well-being.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Finnish Work Environment Fund (Other)
Responsible Party: Principal Investigator, Siiri-Liisi Kraav, Post-doctoral researcher, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240128
Record Dates: First submitted 2024-07-02; First posted 2024-07-11 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Loneliness; Social Isolation; Social Support; Depressive Symptoms
Keywords: loneliness; work well-being; social well-being
MeSH Terms: conditions — Social Isolation; Depression

STUDY DESIGN:
Intervention Model Description: Participants of the intervention group are given access and encouraged to use Frendie PRO mobile application
Masking Description: The baseline data collection is conducted before randomization. No masking will be used after the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Frendie PRO mobile application
- Wait-list controls (No Intervention): The group will have access to the mobile application after the six-month follow-up period.

INTERVENTIONS:
Behavioral: Frendie PRO mobile application — Frendie PRO mobile application offers employees an environment to manage their social relationships, organize leisure activities, and discuss personal or work-related matters.
  Arms: Intervention

SUMMARY:
The goal of this cluster randomized controlled trial is to learn if using Frendie PRO mobile application at workplaces improves social well-being in employees. The main questions it aims to answer are:

Does using Frendie PRO mobile application at work for 6 months reduce loneliness in employees? Does using Fendie PRO mobile application at work for 6 months reduce social isolation in employees?

Researchers will compare employees from workplaces that use the Frendie PRO mobile application to employees from workplaces that do not use the mobile application to see if there are differences in their levels of social well-being (loneliness, social isolation, perceived social support, depressive symptoms).

Participants will be given access to the Frendie PRO mobile application and encouraged to use it by employers.

DETAILED DESCRIPTION:
Participants will be recruited from workplaces that use the Frendie PRO mobile application. After collecting baseline data, each workplace will be randomly assigned to treatment or control conditions. The unit of randomization is a workplace (or a team or department in bigger organizations).

The intervention group will be encouraged to download and start using the Frendie PRO mobile application. The control group will be informed of the date when they will have access to it (six months after the baseline).

Both groups are asked to participate in two follow-ups - a 3-month follow-up and a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All employees working at the company/team/department participating in the study and starting to use the Frendie PRO mobile application within the study period.
* Ability to fill the questionnaires online in Finnish

Exclusion Criteria:

* incapable of using questionnaire online
* does not know Finnish well enough to answer the questions

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1012 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Loneliness | Will be measured three times: baseline, 3-month follow-up and 6-month follow-up
  University of California, Los Angeles (UCLA) Loneliness Scale
Social Isolation | Will be measured three times: baseline, 3-month follow-up and 6-month follow-up
  The Social Isolation scale was modified from an index used by Christiansen et al. (2021). Christiansen and colleagues, in turn, created it inspired by the detailed Social Network Index created by Berkman and Syme (1979).
  Communication frequency with the following groups is measured:
  * family members who live elsewhere
  * friends
  * colleagues or fellow students at the workplace/school and outside of the workplace/school
  * neighbors and local community
  * people from social clubs, hobby groups, and religious organisations at and outside the meetings.

SECONDARY OUTCOMES:
Social support | Will be measured three times: baseline, 3-month follow-up and 6-month follow-up
  Oslo Social Support Scale
Depressive symptoms | Will be measured three times: baseline, 3-month follow-up and 6-month follow-up
  Patient Health Questionnaire-9 (PHQ9)
Workplace loneliness | Will be measured three times: baseline, 3-month follow-up and 6-month follow-up
  Specific scale regarding loneliness experienced at workplaces. Includes 5 items that are modified from the UCLA loneliness scale. It was validated in Finnish adult population. Please see Kemppinen and Tanskanen (2023) for full description:
  Kemppinen, S., Tanskanen, J., 2023. Suomenkielisen työyksinäisyysmittarin validointi etä- ja hybridityöläisillä (Eng title: Validation of Finnish loneliness at work scale with remote and hybrid worker sample). Psykologia 58, 198-219.

OTHER OUTCOMES:
Activity and behavior on the application | 6 months
  Each individual user's activity on the mobile application will be measured. The data will be used for additional analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Siiri-Liisi Kraav, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, North Savonia, Finland

IPD SHARING:
Plan to Share IPD: Yes
After 10 years, anonymized data will be offered to the Finnish Social Science Data Archive. If the data will not be accepted there, it will be destroyed.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After 10 years.
Access Criteria: Application to the Finnish Social Science Data Archive
URL: https://www.fsd.tuni.fi/en/

REFERENCES:
- [Derived] Kraav SL, Schoenmakers E, Linnosmaa I, Sorola S, Tolmunen T. Study protocol of a cluster randomized trial to evaluate the Frendie PRO mobile application's effectiveness in reducing employees' loneliness and social isolation. Contemp Clin Trials. 2025 Oct;157:108060. doi: 10.1016/j.cct.2025.108060. Epub 2025 Aug 28. PMID 40885488